CLINICAL TRIAL: NCT05956145
Title: Effect of Low Dose of Colchicine on Platelet Reactivty in Patients With Chronic Coronary Disease
Brief Title: Effect of Low Dose of Colchicine on Platelet Reactivity
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Sao Paulo (Other)
Responsible Party: Principal Investigator, Jose Carlos Nicolau, Professor, University of Sao Paulo
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: SDC:5007/20/036
Record Dates: First submitted 2022-02-09; First posted 2023-07-21 (Actual); Last update posted 2025-01-17 (Actual); Status verified 2025-01

CONDITIONS: Platelet Aggregation, Spontaneous; Coronary Artery Disease
Keywords: Colchicine; Coronary artery disease; chronic coronary artery disease; inflammation; platelet reactivity
MeSH Terms: conditions — Platelet Aggregation, Spontaneous; Coronary Artery Disease; Inflammation | interventions — Colchicine

STUDY DESIGN:
Intervention Model Description: Prospective, randomized, double-blind, placebo-controlled study.
Who Masked: Participant, Investigator
Masking Description: Double-blind
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention group (Experimental): Colchicine 0.5 mg QD
  Interventions: Drug: Colchicine 0.5 MG
- Placebo group (Placebo Comparator): Placebo
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Colchicine 0.5 MG — Patients with proven chronic coronary disease (documented by a previous history of AMI with or without ST-segment elevation) will be randomized to receive colchicine 0.5 mg once daily (intervention group) or placebo (control group) for a period of 30 ± 3 days.
  Arms: Intervention group
Other: Placebo — Patients with proven chronic coronary disease (documented by a previous history of AMI with or without ST-segment elevation) will be randomized to receive colchicine 0.5 mg once daily (intervention group) or placebo (control group) for a period of 30 ± 3 days.
  Arms: Placebo group

SUMMARY:
Inflammation plays an important role in atherosclerosis and the occurrence of ischemic events. Statins, in addition to their lipid-lowering effect, have also documented anti-inflammatory effect that may partly explain their clinical benefit in reducing cardiovascular ischemic events. Colchicine is an orally administered anti-inflammatory drug that has been used for centuries in several anti-inflammatory or autoimmune diseases. Its mechanism of action occurs by the inhibition of tubulin polymerization and the generation of microtubules and by effects on cell adhesion molecules and inflammatory chemokines. However, there are no studies evaluating the in vivo "antiplatelet action" of colchicine in patients with established cardiovascular disease.

We will evaluate the effect of low-dose 0.5 mg QD colchicine for 30 ± 3 days on platelet reactivity by MultiplateTRAP.

Patients with proven chronic coronary artery disease, that is, documented previous myocardial infarction, will be randomized to receive colchicine 0.5 mg QD or placebo for a period of 30 ± 3 days.

DETAILED DESCRIPTION:
Inflammation plays an important role in atherosclerosis and the occurrence of ischemic events. Statins, in addition to their lipid-lowering effect, have also documented an anti-inflammatory effect that may partly explain their clinical benefit in reducing cardiovascular ischemic events. More recently, canaquinumab, a monoclonal anti-interleukin 1β antibody, significantly reduced vascular events in patients after acute myocardial infarction with residual inflammation, but failed to demonstrate progression to diabetes, including in patients with pre-diabetes. On the other hand, methotrexate has not been shown to be effective in reducing events in a similar population.

In addition to inflammation, thrombosis is directly involved in the pathogenesis of unstable ischemic syndromes. In this context, the association between greater platelet aggregability and clinical events is well established in the literature. The POPULAR study evaluated that after a 1-year follow-up, the primary outcome of death, non-fatal acute myocardial infarction, stent thrombosis or ischemic stroke occurred more frequently in patients with high platelet reactivity undergoing treatment with antiaggregants when evaluated by optical aggregometry and other point of care tests. Another study that evaluated the importance of the platelet response to medications was the ADAPT-DES, in which post-angioplasty patients on dual antiplatelet therapy were at higher risk of complications, especially stent thrombosis, when they presented with high platelet reactivity to clopidogrel. Both studies show the importance of the interaction between platelet changes and the medications that interact in this way and cardiovascular outcomes.

Colchicine is an orally administered anti-inflammatory drug that was initially extracted from autumn saffron and has been used for centuries in various diseases of an anti-inflammatory / autoimmune nature. Its bioavailability after oral administration takes place via uptake in the jejunum and ileum, its lipophilic nature allows it to be absorbed quickly by various types of cells. Its mechanism of action occurs through the inhibition of tubulin polymerization and the generation of microtubules and, possibly, effects on cell adhesion molecules and inflammatory chemokines.

Another route related to colchicine is the suppression of interleukin 1. It is able to prevent the intracellular assembly of the cytosolic protein complex NACHT-LRRPYD 3, responsible for the proteolytic cleavage of caspase-1, which breaks down and activates interleukin 1, blocking its maturation and secretion.

In addition to the action on inflammation, colchicine may be involved in reducing platelet aggregation, as suggested in a mechanistic study that evaluated the in vitro action of colchicine on platelet aggregation in healthy individuals. In this study, in addition to demonstrating the lower aggregability by electrical impedance in the sample subjected to colchicine action, it was found that the drug also exerted effects via inhibition of key proteins involved in the rearrangement of the platelet cytoskeleton. To the best of our knowledge, however, there are no studies evaluating the in vivo "antiplatelet action" of colchicine in patients with established cardiovascular disease.

In the population with coronary heart disease, two important randomized clinical studies have demonstrated the benefit of colchicine: 1) LoDoCo, which demonstrated a reduction in cardiovascular events (composed of infarction, unstable angina, cardiorespiratory arrest or stroke) with a low dose of colchicine in patients with stable coronary disease. ; 2) COLCOT showed a reduction in events, the composite of cardiovascular death, infarction, unstable angina, resuscitated cardiopulmonary arrest or stroke, in patients treated with colchicine after AMI.

Despite the cardiovascular benefit demonstrated in high-risk patients, little is known about the pathophysiological mechanisms involved, being the subject of debates about whether the observed results would be related to the reduction of the progression of atheroscletotic disease, to an antiplatelet effect, or both.

Primary objective: To evaluate the effect of colchicine in low dose for 30 ± 3 days on platelet aggregation by MultiplateTRAP.

Secondary objectives Evaluate the primary objective of the study using Multiplate ADP, ASPI and Collagen.

Exploratory Analysis

Comparison between the colchicine and placebo groups at the end of the 30 ± 3-day follow-up of the following parameters:

* Ultra-sensitive reactive C protein (hs-CRP);
* Interleukin 6 (IL-6);
* Interleukin 1 (IL-1);
* Serum Tromboxane B2;
* Count and fraction of reticulated platelets;
* Mean platelet volume (MPV);
* Total cholesterol / HDL / LDL / triglycerides, apolipoprotein A1, apolipoprotein B;
* Analysis of vascular reactivity;
* Transfer of lipids to HDL.

Analyze the primary outcome of the study in the following subgroups:

* Female versus male;
* Age group ( equal or major to 65 years);
* Presence or not of diabetes mellitus (characterized by use of hypoglycemic drugs previously and / or exam prior to randomization with HbA1c equal or minor to 6.5%);
* LVEF equal or major 40%;
* Obese versus non-obese (BMI equal or major 30)
* Smoker versus non-smoker
* median LDL
* PCRus equal or major 2mg / dl

Study design: Prospective, randomized, double-blind, placebo-controlled study. Patients with proven chronic coronary artery disease, documented by previous history of AMI, will be randomized to receive colchicine 0.5 mg once daily (intervention group) or placebo (control group) for a period of 30 ± 3 days. Randomization will be performed in 2 blocks of 40 patients at a rate of 1: 1. Blood samples will be obtained at the baseline visit and at the end-of-follow-up visit (30 ± 3days after the baseline visit).

Inclusion criteria: Agreement to sign a free and informed consent form; age ≥ 18 years; patients with previous acute myocardial infarction (or more than 1 year according to the criteria of the 4th universal definition using ASA 100mg / day.

Exclusion criteria: Use of any antithrombotic therapy other than AAS for less than 1 week; Stroke in the last 3 months; active infection or current use of systemic antimicrobial therapy; neoplasia in the last 3 years; inflammatory bowel disease or chronic diarrhea; hematological abnormality (Hb ≤ 11g / dL or> 17g / dL, leukocytes ≤ 4,500 / mm3 or> 11,000 / mm3, platelet count <150,000 / mm3 or> 450,000 / mm3); chronic kidney disease (estimated glomerular filtration rate <30 ml / min / 1.73 m2) using the MDRD formula; liver disease defined by CHILD B or C; drug or alcohol abuse; dementia, psychiatric or any condition that, in the researcher's opinion, prevents participation and follow-up in the protocol; history of allergy to colchicine; current treatment with systemic corticosteroids or immunosuppressants.

Sample calculation: In a prior study, published in 2020, it was found an average platelet aggregability by Multiplate-TRAP in patients with chronic coronary disease of 102 AUC +/- 26. Another study analyzing platelet aggregation in vitro in healthy volunteers, found a reduction in aggregability by ADP by 40%. In the present study, for a hypothesis of superiority with a 20% reduction in the mean platelet aggregation in favor of colchicine over placebo, considering an alpha = 0.05 (two-tailed) and a power = 90%, the calculated sample size is 70 patients (35 per group), with a total of 80 being included to compensate for possible losses.

ELIGIBILITY:
Inclusion Criteria:

* Agreement to sign a free and informed consent form (ICF);
* Age equal or major18 years;
* Patients with previous acute myocardial infarction (for more than 1 year) according to the criteria of the 4th universal definition using ASA 100mg / day.

Exclusion Criteria:

* Use of any antithrombotic therapy other than AAS for less than 1 week;
* Stroke in the last 3 months;
* Active infection or current use of systemic antimicrobial therapy;
* Neoplasia in the last 3 years;
* Inflammatory bowel disease or chronic diarrhea;
* Hematological abnormality (Hb equal or minor to11 g / dL or major to17g / dL, Leukocytes minor or equal 4,500 / mm3 or major 11,000 / mm3, platelet count minor 150,000 / mm3 or major450,000 / mm3);
* Chronic kidney disease (estimated glomerular filtration rate <30 ml / min / 1.73 m2) using the MDRD17 formula;
* Liver disease defined by CHILD B or C; 18,19
* Abuse of drugs or alcohol;
* Dementia, psychiatric or any condition that, in the opinion of the researcher, prevents participation and follow-up in the protocol;
* History of allergy to colchicine;
* Current treatment with systemic corticosteroids or immunosuppressants.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2021-06-17 (Actual); Primary Completion 2024-04-03 (Actual); Study Completion 2024-04-03 (Actual)

PRIMARY OUTCOMES:
Platelet aggregation to TRAP | 30 days
  Platelet aggregation assessed by the Multiplate TRAP assay and measured as area under the curve - AUC

SECONDARY OUTCOMES:
Platelet aggregation to ADP | 30 days
  Platelet aggregation assessed by the Multiplate ADP assay and measured as area under the curve - AUC
Platelet aggregation to arachdonic acid | 30 days
  Platelet aggregation assessed by the Multiplate ASPI assay and measured as area under the curve - AUC

OTHER OUTCOMES:
Comparison between the colchicine and placebo groups: | 30 days
  Ultra-sensitive reactive C protein (hs-CRP) ( mg/L )
Comparison between the colchicine and placebo groups: | 30 days
  Interleukin 1 (IL-1)
Comparison between the colchicine and placebo groups: | 30 days
  Interleukin 6 (IL-6)
Comparison between the colchicine and placebo groups: | 30 days
  Count and fraction of reticulated platelets (%)
Comparison between the colchicine and placebo groups: | 30 days
  Cholesterol and fractions in mg/dL
Comparison between the colchicine and placebo groups: | 30 days
  Transfer of lipids to HDL (%)
Comparison between the colchicine and placebo groups: | 30 days
  Average platelet volume (MPV) (fL)

CONTACTS AND LOCATIONS:
Locations (1):
- Heart Institute (InCor) / University of São Paulo, São Paulo, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Hansson GK. Inflammation, atherosclerosis, and coronary artery disease. N Engl J Med. 2005 Apr 21;352(16):1685-95. doi: 10.1056/NEJMra043430. No abstract available. PMID 15843671
- [Background] Ridker PM, Danielson E, Fonseca FA, Genest J, Gotto AM Jr, Kastelein JJ, Koenig W, Libby P, Lorenzatti AJ, MacFadyen JG, Nordestgaard BG, Shepherd J, Willerson JT, Glynn RJ; JUPITER Study Group. Rosuvastatin to prevent vascular events in men and women with elevated C-reactive protein. N Engl J Med. 2008 Nov 20;359(21):2195-207. doi: 10.1056/NEJMoa0807646. Epub 2008 Nov 9. PMID 18997196
- [Background] Ridker PM, Everett BM, Thuren T, MacFadyen JG, Chang WH, Ballantyne C, Fonseca F, Nicolau J, Koenig W, Anker SD, Kastelein JJP, Cornel JH, Pais P, Pella D, Genest J, Cifkova R, Lorenzatti A, Forster T, Kobalava Z, Vida-Simiti L, Flather M, Shimokawa H, Ogawa H, Dellborg M, Rossi PRF, Troquay RPT, Libby P, Glynn RJ; CANTOS Trial Group. Antiinflammatory Therapy with Canakinumab for Atherosclerotic Disease. N Engl J Med. 2017 Sep 21;377(12):1119-1131. doi: 10.1056/NEJMoa1707914. Epub 2017 Aug 27. PMID 28845751
- [Background] Ridker PM, Everett BM, Pradhan A, MacFadyen JG, Solomon DH, Zaharris E, Mam V, Hasan A, Rosenberg Y, Iturriaga E, Gupta M, Tsigoulis M, Verma S, Clearfield M, Libby P, Goldhaber SZ, Seagle R, Ofori C, Saklayen M, Butman S, Singh N, Le May M, Bertrand O, Johnston J, Paynter NP, Glynn RJ; CIRT Investigators. Low-Dose Methotrexate for the Prevention of Atherosclerotic Events. N Engl J Med. 2019 Feb 21;380(8):752-762. doi: 10.1056/NEJMoa1809798. Epub 2018 Nov 10. PMID 30415610
- [Background] Breet NJ, van Werkum JW, Bouman HJ, Kelder JC, Ruven HJ, Bal ET, Deneer VH, Harmsze AM, van der Heyden JA, Rensing BJ, Suttorp MJ, Hackeng CM, ten Berg JM. Comparison of platelet function tests in predicting clinical outcome in patients undergoing coronary stent implantation. JAMA. 2010 Feb 24;303(8):754-62. doi: 10.1001/jama.2010.181. PMID 20179285
- [Background] Stone GW, Witzenbichler B, Weisz G, Rinaldi MJ, Neumann FJ, Metzger DC, Henry TD, Cox DA, Duffy PL, Mazzaferri E, Gurbel PA, Xu K, Parise H, Kirtane AJ, Brodie BR, Mehran R, Stuckey TD; ADAPT-DES Investigators. Platelet reactivity and clinical outcomes after coronary artery implantation of drug-eluting stents (ADAPT-DES): a prospective multicentre registry study. Lancet. 2013 Aug 17;382(9892):614-23. doi: 10.1016/S0140-6736(13)61170-8. Epub 2013 Jul 26. PMID 23890998
- [Background] Imazio M, Brucato A, Cemin R, Ferrua S, Maggiolini S, Beqaraj F, Demarie D, Forno D, Ferro S, Maestroni S, Belli R, Trinchero R, Spodick DH, Adler Y; ICAP Investigators. A randomized trial of colchicine for acute pericarditis. N Engl J Med. 2013 Oct 17;369(16):1522-8. doi: 10.1056/NEJMoa1208536. Epub 2013 Aug 31. PMID 23992557
- [Background] Corps AN, Hesketh TR, Metcalfe JC. Limitations on the use of phenothiazines and local anaesthetics as indicators of calmodulin function in intact cells. FEBS Lett. 1982 Feb 22;138(2):280-4. doi: 10.1016/0014-5793(82)80461-4. No abstract available. PMID 7067838
- [Background] Ravelli RB, Gigant B, Curmi PA, Jourdain I, Lachkar S, Sobel A, Knossow M. Insight into tubulin regulation from a complex with colchicine and a stathmin-like domain. Nature. 2004 Mar 11;428(6979):198-202. doi: 10.1038/nature02393. PMID 15014504
- [Background] Perico N, Ostermann D, Bontempeill M, Morigi M, Amuchastegui CS, Zoja C, Akalin E, Sayegh MH, Remuzzi G. Colchicine interferes with L-selectin and leukocyte function-associated antigen-1 expression on human T lymphocytes and inhibits T cell activation. J Am Soc Nephrol. 1996 Apr;7(4):594-601. doi: 10.1681/ASN.V74594. PMID 8724893
- [Background] Pope RM, Tschopp J. The role of interleukin-1 and the inflammasome in gout: implications for therapy. Arthritis Rheum. 2007 Oct;56(10):3183-8. doi: 10.1002/art.22938. No abstract available. PMID 17907163
- [Background] Martinon F, Petrilli V, Mayor A, Tardivel A, Tschopp J. Gout-associated uric acid crystals activate the NALP3 inflammasome. Nature. 2006 Mar 9;440(7081):237-41. doi: 10.1038/nature04516. Epub 2006 Jan 11. PMID 16407889
- [Background] Niel E, Scherrmann JM. Colchicine today. Joint Bone Spine. 2006 Dec;73(6):672-8. doi: 10.1016/j.jbspin.2006.03.006. Epub 2006 Sep 1. PMID 17067838
- [Background] Cimmino G, Tarallo R, Conte S, Morello A, Pellegrino G, Loffredo FS, Cali G, De Luca N, Golino P, Trimarco B, Cirillo P. Colchicine reduces platelet aggregation by modulating cytoskeleton rearrangement via inhibition of cofilin and LIM domain kinase 1. Vascul Pharmacol. 2018 Dec;111:62-70. doi: 10.1016/j.vph.2018.09.004. Epub 2018 Oct 1. PMID 30287213
- [Background] Nidorf SM, Eikelboom JW, Budgeon CA, Thompson PL. Low-dose colchicine for secondary prevention of cardiovascular disease. J Am Coll Cardiol. 2013 Jan 29;61(4):404-410. doi: 10.1016/j.jacc.2012.10.027. Epub 2012 Dec 19. PMID 23265346
- [Background] Tardif JC, Kouz S, Waters DD, Bertrand OF, Diaz R, Maggioni AP, Pinto FJ, Ibrahim R, Gamra H, Kiwan GS, Berry C, Lopez-Sendon J, Ostadal P, Koenig W, Angoulvant D, Gregoire JC, Lavoie MA, Dube MP, Rhainds D, Provencher M, Blondeau L, Orfanos A, L'Allier PL, Guertin MC, Roubille F. Efficacy and Safety of Low-Dose Colchicine after Myocardial Infarction. N Engl J Med. 2019 Dec 26;381(26):2497-2505. doi: 10.1056/NEJMoa1912388. Epub 2019 Nov 16. PMID 31733140
- [Background] Thygesen K, Alpert JS, Jaffe AS, Chaitman BR, Bax JJ, Morrow DA, White HD; Executive Group on behalf of the Joint European Society of Cardiology (ESC)/American College of Cardiology (ACC)/American Heart Association (AHA)/World Heart Federation (WHF) Task Force for the Universal Definition of Myocardial Infarction. Fourth Universal Definition of Myocardial Infarction (2018). Circulation. 2018 Nov 13;138(20):e618-e651. doi: 10.1161/CIR.0000000000000617. No abstract available. PMID 30571511
- [Background] Levey AS, Bosch JP, Lewis JB, Greene T, Rogers N, Roth D. A more accurate method to estimate glomerular filtration rate from serum creatinine: a new prediction equation. Modification of Diet in Renal Disease Study Group. Ann Intern Med. 1999 Mar 16;130(6):461-70. doi: 10.7326/0003-4819-130-6-199903160-00002. PMID 10075613
- [Background] Child CG, Turcotte JG. Surgery and portal hypertension. Major Probl Clin Surg. 1964;1:1-85. No abstract available. PMID 4950264
- [Background] Pugh RN, Murray-Lyon IM, Dawson JL, Pietroni MC, Williams R. Transection of the oesophagus for bleeding oesophageal varices. Br J Surg. 1973 Aug;60(8):646-9. doi: 10.1002/bjs.1800600817. No abstract available. PMID 4541913
- [Background] Arantes FBB, Menezes FR, Franci A, Barbosa CJDG, Dalcoquio TF, Nakashima CAK, Baracioli LM, Furtado RHM, Nomelini QSS, Ramires JAF, Kalil Filho R, Nicolau JC. Influence of Direct Thrombin Inhibitor and Low Molecular Weight Heparin on Platelet Function in Patients with Coronary Artery Disease: A Prospective Interventional Trial. Adv Ther. 2020 Jan;37(1):420-430. doi: 10.1007/s12325-019-01153-8. Epub 2019 Nov 22. PMID 31758517
- [Background] von Pape KW, Dzijan-Horn M, Bohner J, Spannagl M, Weisser H, Calatzis A. [Control of aspirin effect in chronic cardiovascular patients using two whole blood platelet function assays. PFA-100 and Multiplate]. Hamostaseologie. 2007 Aug;27(3):155-60; quiz 161-2. doi: 10.1007/978-3-540-36715-4_49. German. PMID 17694222
- [Background] Sibbing D, Braun S, Jawansky S, Vogt W, Mehilli J, Schomig A, Kastrati A, von Beckerath N. Assessment of ADP-induced platelet aggregation with light transmission aggregometry and multiple electrode platelet aggregometry before and after clopidogrel treatment. Thromb Haemost. 2008 Jan;99(1):121-6. doi: 10.1160/TH07-07-0478. PMID 18217143
- [Background] Lo Prete AC, Dina CH, Azevedo CH, Puk CG, Lopes NH, Hueb WA, Maranhao RC. In vitro simultaneous transfer of lipids to HDL in coronary artery disease and in statin treatment. Lipids. 2009 Oct;44(10):917-24. doi: 10.1007/s11745-009-3342-2. Epub 2009 Sep 16. PMID 19760244
- [Background] Kuvin JT, Patel AR, Sliney KA, Pandian NG, Sheffy J, Schnall RP, Karas RH, Udelson JE. Assessment of peripheral vascular endothelial function with finger arterial pulse wave amplitude. Am Heart J. 2003 Jul;146(1):168-74. doi: 10.1016/S0002-8703(03)00094-2. PMID 12851627
- [Background] Hamburg NM, Benjamin EJ. Assessment of endothelial function using digital pulse amplitude tonometry. Trends Cardiovasc Med. 2009 Jan;19(1):6-11. doi: 10.1016/j.tcm.2009.03.001. PMID 19467447